CLINICAL TRIAL: NCT02516982
Title: Tablet Computers for Implementing NICE Antenatal Mental Health Guidelines - Feasibility Study
Brief Title: mHealth for Antenatal Mental Health
Acronym: AMHS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15IC2687
Record Dates: First submitted 2015-07-20; First posted 2015-08-06 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Depression; Pregnancy
Keywords: mHealth; Telemedicine; Perinatal depression; Screening; Edinburgh Postnatal Depression Scale; Whooley Questions; Data collection; Mood disorders; Mental health; Antenatal care; Prenatal Care
MeSH Terms: conditions — Depression; Mood Disorders; Psychological Well-Being | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Screening - Scrolling layout: Participants will be asked to complete a survey consisting of three sections using an iPad Air tablet:
  * Section 1: Demographic information survey
  * Section 2: Whooley questions
  * Section 3: Edinburgh Postnatal Depression Scale
  All questions will be presented on a single screen. This means that participants will have to scroll vertically in order to answer all the questions.
  Interventions: Other: Whooley Questions; Other: Edinburgh Postnatal Depression Scale
- Screening - Paging layout: Participants will be asked to complete a survey consisting of three sections using an iPad Air tablet:
  * Section 1: Demographic information survey
  * Section 2: Whooley questions
  * Section 3: Edinburgh Postnatal Depression Scale
  Only one question will be presented at any given time. This means that participants will have to navigate through multiple pages in order to answer all the questions.
  Interventions: Other: Whooley Questions; Other: Edinburgh Postnatal Depression Scale
- Retrospective plus momentary assessment: Participants in this group will be asked to download and install an app onto their own smartphones. After that, they will be asked to complete a sampling protocol consisting of 6 consecutive days, once a month for 6 months. During the 6 assessment days, participants will be required to complete the Edinburgh Postnatal Depression Scale, 5 momentary questions on a 5-point pictorial scale, and 2 contextual questions.
  Interventions: Other: Edinburgh Postnatal Depression Scale; Other: Momentary questions; Other: Contextual questions
- Retrospective assessment: Participants in this group will be asked to download and install an app onto their own smartphones. After that, they will be asked to complete a sampling protocol consisting of one day a month for 6 months. The assessment days will consist of a single administration of the Edinburgh Postnatal Depression Scale.
  Interventions: Other: Edinburgh Postnatal Depression Scale

INTERVENTIONS:
Other: Whooley Questions — The Whooley questions are a case-finding instrument for depression in primary care. This 2-question instrument screens for depressed mood and anhedonia that have been present during the past month. Respondents are required to answer Yes or No to each of these questions. An affirmative answer to any of them should be followed by further assessment, including the use of a validated screening instrument or referral to a general practitioner or a mental health practitioner.
  Groups: Screening - Paging layout; Screening - Scrolling layout
Other: Edinburgh Postnatal Depression Scale — The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-administered survey that screens for symptoms such as feelings of guilt, sleep disturbance, reduced energy levels, anhedonia and suicidal ideation that have been present during the 7 days preceding its administration. Each question is scored on a 4-point scale ranging from 0 to 3 points. Overall scores between 10 and 12 points suggest increased risk for depression; scores of 13 points or above indicate that the diagnostic criteria for major depression disorder have probably been met. In addition, item 10 deals with suicidal thoughts. The EPDS is a valid and reliable tool for identifying women at risk of depression, both during pregnancy and postpartum, and is sensitive to changes in the severity of depression over time.
Other: Momentary questions — These will consist of 5 questions on a 5-point pictorial scales, assessing participants' mood, sleep, energy, enjoyment and worry.
  Groups: Retrospective plus momentary assessment
Other: Contextual questions — Two questions asking for participants' location and activity at the time they were asked to complete the momentary questions.
  Groups: Retrospective plus momentary assessment

SUMMARY:
The aim of this study is to determine the feasibility of using mobile technology for:

1. Implementing the recommendations of the Antenatal and postnatal mental health: clinical management and service guidance NICE guideline for recognising depression (i.e., Whooley questions followed by a validated screening instrument such as the Edinburgh Postnatal Depression Scale) during pregnancy using iPad Air tablets in the waiting area of general practices, midwifery services, or hospitals during antenatal clinics; and
2. Using a bespoke app running on pregnant women's own smartphones to monitor mood and symptoms of depression throughout pregnancy.

DETAILED DESCRIPTION:
As part of our first aim, we will assess the psychometric properties of the Whooley questions, by comparing the answers given to these questions against the scores obtained on the Edinburgh Postnatal Depression Scale, and we will manipulate the survey questionnaire layout of the Whooley Questions and the Edinburgh Postnatal Depression Scale in order to ensure that this survey design choice does not affect data quality. As part of our second aim, we will compare two prospective sampling protocols on patient compliance and engagement with the app.

We will use a parallel, randomised control trial study design. Participation in each part of the study (i.e., iPads in antenatal clinics, or app running on own handset) will be independent from each other. Those participants consenting to get involved in the part of the study assessing the use of iPads in antenatal clinics will be randomly assigned to complete (i) an app version of the Whooley questions and the Edinburgh Postnatal Depression Scale in which the questionnaires are presented using a scrolling layout (i.e., App screening - Scrolling), or (ii) an app version of the Whooley questions and the Edinburgh Postnatal Depression Scale in which the questionnaires are presented using a paging layout (i.e., App screening - Paging).

Participants consenting to get involved in the part of the study assessing the use of an app running on participants' own devices will be randomly allocated to one of two sampling protocols: (i) a prospective sampling protocol of 6 months consisting of the Edinburgh Postnatal Depression Scale and 5 momentary questions related to mood; or (ii) a prospective sampling protocol of 6 months consisting of the Edinburgh Postnatal Depression Scale.

We will utilise a block randomisation procedure (with blocks of 4) to generate our allocation sequence. Random numbers will be generated using Stata 13.0. Researchers conducting participant recruitment will not be involved in this randomisation procedure in order to avoid recruitment bias.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal clinics

Exclusion Criteria:

* Diagnosis of any common mental health disorder (i.e., depression or anxiety disorders) as specified in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition
* Receiving treatment for any common mental health disorder
* Recent personal history of any common mental health disorder (i.e., within the past 12 months)
* Not comfortable reading and writing in English

Participants enrolled in the study assessing an app for the monitoring of mood and symptoms of depression need to own an iPhone or any Android-compatible smartphone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are 18 years old or older.
Sampling Method: Probability Sample
Enrollment: 946 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose S Marcano Belisario, Principal Investigator — Imperial College London; Josip Car, Principal Investigator — Imperial College London; Cecily Morrison, Principal Investigator — Imperial College London; John O'Donoghue, Principal Investigator — Imperial College London; Ajay Gupta, Study Chair — Imperial College London; Paul Ramchandani, Study Chair — Imperial College London; Gavin Doherty, Principal Investigator — University of Dublin, Trinity College; Kevin Doherty, Principal Investigator — University of Dublin, Trinity College
Locations (14):
- United Kingdom (14):
  - East Lancashire, Blackburn
  - Royal Bolton Hospital, Bolton
  - Burton Hospitals, Burton
  - The Pennine Acute Hospitals, Crumpsall
  - Hinchinbrooke Hospital, Huntingdon
  - East Midlands CRN, Lincoln
  - Chelsea & Westminster Hospital, London
  - Hillingdon Hospitals, London
  - Northwick Park Hospital, London
  - West Middlesex Hospital, London
  - North of England, Newcastle
  - Shrewsburty & Telford Hospital, Shrewsbury
  - University Hospitals of North Midlands, Stoke-on-Trent
  - Wrightington, Wigan and Leigh NHS, Wigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marcano-Belisario JS, Gupta AK, O'Donoghue J, Morrison C, Car J. Tablet computers for implementing NICE antenatal mental health guidelines: protocol of a feasibility study. BMJ Open. 2016 Jan 22;6(1):e009930. doi: 10.1136/bmjopen-2015-009930. PMID 26801468
- [Background] Marcano Belisario JS, Doherty K, O'Donoghue J, Ramchandani P, Majeed A, Doherty G, Morrison C, Car J. A bespoke mobile application for the longitudinal assessment of depression and mood during pregnancy: protocol of a feasibility study. BMJ Open. 2017 May 29;7(5):e014469. doi: 10.1136/bmjopen-2016-014469. PMID 28554914
- [Result] Marcano-Belisario JS, Gupta AK, O'Donoghue J, Ramchandani P, Morrison C, Car J. Implementation of depression screening in antenatal clinics through tablet computers: results of a feasibility study. BMC Med Inform Decis Mak. 2017 May 10;17(1):59. doi: 10.1186/s12911-017-0459-8. PMID 28490353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1: Scrolling vs Paging layouts - Recruitment dates: October 2015 to May 2016 Phase 2: Momentary vs Momentary plus Retrospective - Recruitment dates: April 2017 tp August 2017
Groups:
- Screening - Scrolling Layout: Participants were asked to complete the following surveys using an iPad in the waiting area of antenatal clinics: Demographic information survey; Whooley questions; and the Edinburgh Postnatal Depression Scale.
  All questions were presented on a single screen. This means that participants had to scroll vertically to answer all the questions.
- Screening - Paging Layout: Participants were asked to complete the following surveys using an iPad in the waiting area of antenatal clinics: Demographic information survey; Whooley questions; and the Edinburgh Postnatal Depression Scale.
  Only one question was displayed on the screen at any given time. This means that participants had to navigate through multiple pages in order to answer all the questions.
- Retrospective Plus Momentary Assessment: Participants in this group were asked to download and install an app onto their own smartphones. After that, they were be asked to complete a sampling protocol consisting of 6 consecutive days, once a month for 6 months. During the 6 assessment days, participants were required to complete the Edinburgh Postnatal Depression Scale, 5 momentary questions on a 5-point pictorial scale, and 2 contextual questions.
- Retrospective Assessment: Participants in this group were asked to download and install an app onto their own smartphones. After that, they were asked to complete a sampling protocol consisting of one day a month for 6 months. The assessment days consisted of a single administration of the Edinburgh Postnatal Depression Scale.
Period: Overall Study
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout | Retrospective Plus Momentary Assessment | Retrospective Assessment
Started | 305 | 292 | 174 | 175
Completed | 273 | 257 | 126 | 125
Not Completed | 32 | 35 | 48 | 50
Not completed — Called in to antenatal appointment | 32 | 35 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Did not install the app | 0 | 0 | 46 | 47

BASELINE CHARACTERISTICS:
Groups:
- Screening - Scrolling Layout: Participants were asked to complete the following surveys using an iPad in the waiting area of antenatal clinics: Demographic information survey; Whooley questions; and Edinburgh Postnatal Depression Scale.
  All questions were presented on a single screen. This means that participants had to scroll vertically to answer all the questions.
- Screening - Paging Layout: Participants were asked to complete the following surveys using an iPad in the waiting area of antenatal clinics: Demographic information survey; Whooley questions; and Edinburgh Postnatal Depression Scale.
  Only one question was displayed on the screen at any given time. This means that participants had to navigate through multiple pages in order to answer all the questions.
- Retrospective Plus Momentary Assessment: Participants in this group were asked to download and install an app onto their own smartphones. After that, they were asked to complete a sampling protocol consisting of 6 consecutive days, once a month for 6 months. During the 6 assessment days, participants were required to complete the Edinburgh Postnatal Depression Scale, 5 momentary questions on a 5-point pictorial scale, and 2 contextual questions.
- Total: Total of all reporting groups
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout | Retrospective Plus Momentary Assessment | Retrospective Assessment | Total
Number analyzed (Participants) | 305 | 292 | 174 | 175 | 946
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18 - 22 years | 23 | 19 | 17 | 10 | 69
  Age group: 23 - 27 years | 51 | 45 | 32 | 46 | 174
  Age group: 28 - 32 years | 108 | 113 | 57 | 63 | 341
  Age group: 33 - 37 years | 87 | 85 | 49 | 44 | 265
  Age group: 38+ years | 36 | 30 | 19 | 12 | 97
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 305 | 292 | 174 | 175 | 946
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnich background: White | 179 | 190 | 146 | 153 | 668
  Ethnich background: Mixed | 15 | 13 | 3 | 1 | 32
  Ethnich background: Asian | 70 | 51 | 16 | 15 | 152
  Ethnich background: Black | 20 | 21 | 0 | 0 | 41
  Ethnich background: Other | 18 | 17 | 6 | 6 | 47
  Ethnich background: Not disclosed | 3 | 0 | 3 | 0 | 6
Relationship status [Count of Participants; unit: Participants]
  Single | 24 | 21 | 36 | 43 | 124
  Married/civil partnership | 201 | 187 | 126 | 116 | 630
  Cohabiting | 74 | 72 | 0 | 0 | 146
  Divorced/widowed/separated | 3 | 7 | 2 | 2 | 14
  Not disclosed | 3 | 5 | 10 | 14 | 32
Employment status [Count of Participants; unit: Participants]
  Full-time employment | 141 | 148 | 93 | 82 | 464
  Part-time employment | 58 | 54 | 38 | 40 | 190
  Self-employed | 30 | 26 | 16 | 22 | 94
  Seeking employment | 11 | 19 | 3 | 8 | 41
  Unemployed | 54 | 39 | 24 | 23 | 140
  Disability | 11 | 6 | 0 | 0 | 17
Highest educational achievement [Count of Participants; unit: Participants]
  Postgraduate degree | 56 | 53 | 0 | 0 | 109
  University degree | 124 | 112 | 93 | 100 | 429
  College degree or below | 108 | 110 | 31 | 33 | 282
  None | 8 | 6 | 1 | 8 | 23
  Other qualification | 9 | 11 | 49 | 34 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Responding Affirmatively to at Least One Whooley Question According to Survey Layout
Description: Comparison of the number of participants answering affirmatively to at least one Whooley question in each experimental group. This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups.
Time Frame: One-off assessment immediately after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Participants | 62 | 60
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.994, Chi-squared, Corrected

2. Primary Outcome: Median EPDS Scores According to Survey Layout
Description: This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups. Median scores on the Edinburgh Postnatal Depression Scale according to group allocation. The EPDS consists of 10 questions each rated on a 4-point scale ranging from 0 to 3 points. Overall scores are obtained by adding the scores of all the individual questions, and range from 0 points to 30 points. Overall scores of 0 to 9 points suggest a low risk of perinatal depression. Overall scores between 10 and 12 points suggest an increased risk of perinatal depression. Overall scores of 13 points or more suggest that the respondent is likely to have met the diagnostic criteria for perinatal depression. Moreover, scores of 1 point or more on question 10 of the EPDS ought to be explored further as this question deals with ideas of self-harm.
Time Frame: One-off assessment immediately after recruitment
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Score on a scale | 3 [0 to 21] | 3 [0 to 17]
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Participants at Each EPDS Scoring Interval According to Survey Layout
Description: Number of participants scoring at each of the scoring intervals that have been reported for the Edinburgh Postnatal Depression Scale: 0 to 9 points - low risk; 10 to 12 points - moderate risk; 13 points or more - high risk. This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups.
Time Frame: One-off assessment immediately after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Participants
  0 - 9 points | 236 | 225
  10 - 12 points | 14 | 24
  13+ points | 23 | 8
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.008, Chi-squared, Corrected

4. Primary Outcome: Number of Participants According to Their Score on Question 10 of the EPDS According to Survey Layout
Description: Number of participants scoring 1 point or more on question 10 of the Edinburgh Postnatal Depression Scale, which deals with thoughts of self-harm. This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups.
Time Frame: One-off assessment immediately after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Participants
  0 points | 268 | 251
  1+ points | 5 | 6
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.919, Chi-squared, Corrected

5. Primary Outcome: Adherence With a 6-month Follow-up Protocol
Description: This outcome was measured on the retrospective plus momentary assessment and retrospective assessment groups only. Participants who completed at least one expected assessment during each sampling period
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Plus Momentary Assessment | Retrospective Assessment
Number analyzed (Participants) | 174 | 175
Participants | 22 | 3
Statistical Analysis 1: Comparison: Retrospective Plus Momentary Assessment vs Retrospective Assessment; Test type: Superiority; p = 0.0001467, Chi-squared, Corrected

6. Secondary Outcome: Time Needed to Complete the Whooley Questions and the EPDS According to Survey Layout
Description: This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups. Time elapsed (in seconds) between the participants starting to read the basic instructions on how to complete the survey questionnaires and the participant completing the EPDS. These actions will be indicated by participants pressing the Start button on the device screen and when a message acknowledging that they have completed the survey questionnaires is displayed on the device screen. This component will be broken down further into the individual survey questionnaires that participants will be required to complete (i.e., personal demographic information, Whooley questions, and EPDS). In addition, we will account for the time that participants spend experiencing problems, distractions or making requests for help or clarification.
Time Frame: One-off assessment immediately after recruitment
Measure: Median (Full Range); unit: Seconds
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Seconds | 285.5 [107 to 3444] | 333 [135 to 3146]
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Proportion of Participants Requesting Technical Assistance According to Survey Layout
Description: This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups. Number of participants who made no requests for technical assistance, and those who requested technical assistance
Time Frame: One-off assessment immediately after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Participants
  No requests | 254 | 241
  Requests made | 19 | 16
Statistical Analysis 1: Comparison: Screening - Scrolling Layout vs Screening - Paging Layout; Test type: Superiority; p = 0.869, Chi-squared, Corrected

8. Secondary Outcome: Number of Requests for Technical Assistance by Type of Request and According to Survey Layout
Description: This outcome was only measured in the Screening - Scrolling layout and in the Screening - Paging layout groups. Total number of requests for technical assistance made in each experimental group according to type of request.
Time Frame: One-off outcome assessment conducted up to 24 hours after obtaining written, informed consent
Measure: Number; unit: Requests for technical assistance
Units Other Than Participants: Requests for technical assistance
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout
Number analyzed (Participants) | 273 | 257
Number analyzed (Requests for technical assistance) | 19 | 16
Requests for technical assistance
  Clarification of questions | 14 | 11
  Interface issues | 1 | 1
  Navigation issues | 0 | 3
  Not recorded | 4 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants did not receive a medical intervention. Therefore, no mortality or serious adverse events were expected in this trial. We defined adverse events as those pregnant women who scored above the recommended threshold for the EPDS (i.e., 13 points or more) and had to be referred to specialist mental health services as a result of this.
Arm/Group | Screening - Scrolling Layout | Screening - Paging Layout | Retrospective Plus Momentary Assessment | Retrospective Assessment
All-Cause Mortality (participants affected / at risk) | 0/273 | 0/257 | 0/174 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/273 | 0/257 | 0/174 | 0/175
Other Adverse Events (participants affected / at risk) | 23/273 | 8/257 | 25/174 | 26/175
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Screening - Scrolling Layout (N=273) | Screening - Paging Layout (N=257) | Retrospective Plus Momentary Assessment (N=174) | Retrospective Assessment (N=175)
Thirteen points or more on the EPDS at baseline (Psychiatric disorders) | 23 (23) | 8 (8) | 6 (6) | 9 (9) — Scoring 13 points or more on the EPDS
Thirteen points or more on the EPDS during a six-month follow up (Psychiatric disorders) | 0/0 (0) | 0/0 (0) | 25 (37) | 26 (51) — Scoring 13 points or more on the EPDS at any point during 6 month follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02516982/Prot_SAP_000.pdf